CLINICAL TRIAL: NCT07153133
Title: Efficacy of Albumin Platelet Rich Fibrin on Complications After Mandibular Third Molar Extraction: A Clinical and Biochemical Study
Brief Title: Efficacy of Albumin Platelet Rich Fibrin on Complications After Mandibular Third Molar Extraction.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nader Matrouk Farag AL-Saihani, Clinical Demonstrator at oral and maxillofacial surgery department, Faculty of dentistry, Mansoura University, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ms.25.03.5
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-03

CONDITIONS: Tooth Extraction Site Healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): sixteen teeth extraction socket left for normal healing (blood Clot)
- study group (Experimental): sixteen teeth extraction socket filled by albumin platelet rich fibrin
  Interventions: Biological: albumin platelet rich fibrin

INTERVENTIONS:
Biological: albumin platelet rich fibrin — sixteen teeth extraction socket filled by albumin platelet rich fibrin
  Arms: study group

SUMMARY:
Sixteen patients with bilateral impacted lower third molars seeking treatment will be recruited from the out-patient clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry at Mansoura University.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients classified as ASA (American Society of Anesthesiologists) Physical Status Classification Class I.
* Patients seeking extraction of both mandibular third molars.
* Patients aged 18 - 40 years old by the day of surgery.
* Patients willing to participate in the study and commit to regular follow-up appointments.

Exclusion Criteria:

* Heavy Smokers (more than 25 cigarettes per day).
* Patients with Poor oral hygiene.
* Patients with history of a chemotherapy or radiotherapy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Facial Swelling (Edema) | first day, third day and seventh day after surgery
  Swelling will be evaluated using a tape measure with three measurements performed on the patient's operated site using five reference points:
  * A) Lateral corner of the eye/angle of the mandible
  * B) Tragus/outer corner of the mouth
  * C) Tragus/soft tissue pogonion
  * Measurements will be taken before surgery (baseline). Swelling will be evaluated by comparing the difference between preoperative and postoperative measurements.
Wound Healing | first day, third day and seventh day
  The area of operation will be examined for signs and symptoms of infection, including: swelling, redness, hotness, pus discharge.
  * Any manifestations of wound healing disturbance, including:
  * Wound dehiscence
  * Exposure of underlying hard tissue will be carefully noted
3- Postoperative pain severity | first day, third day and seventh day
  Pain will be evaluated using Visual Analogue Scale (VAS) which is a 10- points (cm) scale, in which the minimum end '0" represents no pain, while the maximum end 10" represents the worst pain. Patients, after being informed about the VAS by the operator, identified the VAS score and the operator recorded them in their charts.
4- blood test | first day, third day and seventh day
  1. 5 cm of blood will be withdrawn under aseptic conditions using sterile venipuncture.
  2. Blood will be separated immediately by centrifugation (3000 rpm).
  3. Serum samples will be frozen at -20°C until assay.
  4. Serum concentrations of interleukin 6, macrophage inflammatory protein, granulocyte macrophage colony-stimulation factor, and vascular endothelial growth factor will be assessed using enzyme-linked immunosorbent assays (ELISA) kits according to the manufacturer's protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura Universty, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided